CLINICAL TRIAL: NCT00736879
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled, Parallel Group, Phase III Trial to Evaluate the Safety and Efficacy of Dapagliflozin as Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet and Exercise
Brief Title: Safety and Efficacy of Dapagliflozin as Monotherapy in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-032
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dapagliflozin 1 mg (Experimental): Dapagliflozin: 1 mg
  Interventions: Drug: Dapagliflozin
- Dapagliflozin 2.5 mg (Experimental): Dapagliflozin: 2.5 mg
  Interventions: Drug: Dapagliflozin
- Dapagliflozin 5 mg (Experimental): Dapagliflozin: 5 mg
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo: 0 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, Once Daily, Up to 24 weeks
  Other Names: BMS-512148; Farxiga™
  Arms: Dapagliflozin 1 mg; Dapagliflozin 2.5 mg; Dapagliflozin 5 mg
Drug: Placebo — Tablets, Oral, Once Daily, Up to 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this clinical research study is to learn if BMS-512148 (Dapagliflozin) can help reduce the blood sugar levels in subjects with Type 2 Diabetes who are not well controlled on diet and exercise alone. The safety of this treatment will also be studied

ELIGIBILITY:
Inclusion Criteria:

* Male and females, ≥18 to ≤77 years old, with type 2 diabetes mellitus
* Subjects must have central laboratory pre-randomization A1C ≥7.0 and ≤ 10.0%
* C-peptide ≥ 1.0 ng/mL (0.34 nmol/L)
* Body Mass Index ≤ 45 kg/m²
* Must be able to perform self monitoring of blood glucose

Exclusion Criteria:

* aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3* upper limit of normal (ULN)
* Serum Total bilirubin >2 mg/dL (34.2 µmol/L)
* Creatinine kinase >3* ULN
* Serum creatinine ≥1.50 mg/dL (133 µmol/L) for male subjects, ≥1.40 mg/dL (124 µmol/L) for female subjects
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncological, endocrine, psychiatric, or rheumatic diseases

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2008-09-22 (Actual); Primary Completion 2009-12-29 (Actual); Study Completion 2009-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (55):
- United States (26):
  - Dedicated Clinical Research, Litchfield Park, Arizona
  - 43rd Medical Associates, P.C., Phoenix, Arizona
  - Clinical Research Advantage, Inc., Tempe, Arizona
  - Valley Research, Fresno, California
  - Marina Raikhel, Md, Faafp, Lomita, California
  - Richard S. Cherlin, Md, Los Gatos, California
  - Orange County Research Center, Tustin, California
  - Family Physicians Of Greeley, Greeley, Colorado
  - Coastal Connecticut Research, Llc, New London, Connecticut
  - Central Florida Clinical Trials, Inc., Altamonte Springs, Florida
  - Westside Center For Clinical Research, Jacksonville, Florida
  - Panhandle Family Care Associates, Marianna, Florida
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Belzoni Clinical Research, Belzoni, Mississippi
  - R-Research, Hamilton, New Jersey
  - Internist Associates Of Central New York, Syracuse, New York
  - Southgate Medical Group, West Seneca, New York
  - Down East Medical Associates, Pa, Morehead City, North Carolina
  - James J. Brown, Md, Akron, Ohio
  - Integris Family Care South, Oklahoma City, Oklahoma
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - Abbott Clinical Research Group, Inc, San Antonio, Texas
  - Avastra Clinical Trials, Midvale, Utah
  - Optimum Clinical Research, Inc., Salt Lake City, Utah
  - Capital Clinical Research Center, Olympia, Washington
  - Stephen G. Danley, Do, Spokane, Washington
- Canada (10):
  - Local Institution, Calgary, Alberta
  - Local Institution, Coquitlam, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, Ajax, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Waterloo, Ontario
  - Local Institution, Drummondville, Quebec
  - Local Institution, L'Ancienne-Lorette, Quebec
  - Local Institution, Saint-Léonard, Quebec
- India (3):
  - Local Institution, Ahmedabad
  - Local Institution, Bangalore
  - Local Institution, Jaipur
- Mexico (7):
  - Local Institution, Durango, Durango
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Veracruz, Veracruz
  - Local Institution, Mérida, Yucatán
- Local Institution, Ponce, Puerto Rico
- Russia (4):
  - Local Institution, Kursk
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Smolensk
- South Africa (4):
  - Local Institution, Benoni, Gauteng
  - Local Institution, Soweto, Gauteng
  - Local Institution, Paarl, Western Cape
  - Local Institution, Tygerberg, Western Cape

REFERENCES:
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated 22 September 2008 and completed 29 December 2009 in drug naive participants with type 2 diabetes mellitus who had inadequate glycemic control, defined as an hemoglobin A1c (HbA1c) greater than, equal to ( ≥) 7.0% and less than equal to (≤) 10.0%, with diet and exercise.
Pre-assignment Details: 497 enrolled in Qualification Period: 297 completed: 13 withdrew consent, 1 lost to follow up (LTF), 1 pregnancy, 183 no longer met criteria, 2 other; 297 entered Placebo Lead-In Period: 282 completed: 3 withdrew consent, 4 LTF, 5 no longer met criteria, 3 other. 282 treated Double Blind; Follow Up visit: 4 weeks ± 5 days post treatment completion.
Groups:
- Placebo: Placebo tablets matching either 1 mg, 2.5 mg, or 5 mg dapagliflozin tablets were taken orally once daily (with morning meal) for 24 weeks during the Double Blind Treatment Period.
- Dapagliflozin 1mg: 1 mg dapagliflozin tablets were taken orally once daily (with morning meal) for 24 weeks during the Double Blind Treatment Period.
- Dapagliflozin 2.5 mg: 2.5 mg dapagliflozin tablets were taken orally once daily (with morning meal) for 24 weeks during the Double Blind Treatment Period.
- Dapagliflozin 5 mg: 5 mg dapagliflozin tablets were taken orally once daily (with morning meal) for 24 weeks during the Double Blind Treatment Period.
Period: Double Blind Treatment Period
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Started | 68 | 72 | 74 | 68
Completed | 65 | 68 | 67 | 63
Not Completed | 3 | 4 | 7 | 5
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Poor non-compliance | 0 | 0 | 1 | 1
Not completed — No longer met criteria | 0 | 1 | 0 | 0
Not completed — non-specified | 0 | 1 | 0 | 0
Period: Follow up Period - No Drug Treatment
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Started | 66 (Those not completing 24 weeks of treatment can still remain in the trial for 4 weeks of follow up.) | 70 (Those not completing 24 weeks of treatment can still remain in the trial for 4 weeks of follow up.) | 66 (Those not completing 24 weeks of treatment can still remain in the trial for 4 weeks of follow up.) | 62 (Those not completing 24 weeks of treatment can still remain in the trial for 4 weeks of follow up.)
Completed | 65 | 67 | 66 | 62
Not Completed | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — non-specified | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who took at least one dose of double-blind study medication were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Total
Number analyzed (Participants) | 68 | 72 | 74 | 68 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (11.08) | 53.7 (9.04) | 53.5 (10.61) | 51.3 (11.51) | 53.0 (10.57)
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 55 | 63 | 61 | 61 | 240
  Greater than, equal to (>=) 65 and < 75 years | 11 | 9 | 12 | 6 | 38
  >= 75 years | 2 | 0 | 1 | 1 | 4
  Not Reported | 0 | 0 | 0 | 0 | 0
Age, Customized [Number; unit: participants] — Female age less than equal to (<=) 50 years and greater than (>) 50 years.
  participants
    Female <= 50 years | 10 | 12 | 11 | 22 | 55
    Female > 50 years | 21 | 22 | 29 | 14 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 40 | 36 | 141
  Male | 37 | 38 | 34 | 32 | 141
Race/Ethnicity, Customized [Number; unit: participants]
  White | 57 | 56 | 61 | 55 | 229
  Black/African American | 3 | 4 | 2 | 3 | 12
  Asian | 7 | 11 | 10 | 10 | 38
  Other Race | 1 | 1 | 1 | 0 | 3
  Ethnicity Hispanic/Latino | 3 | 1 | 2 | 3 | 9
  Ethnicity Not Hispanic/Latino | 10 | 13 | 11 | 9 | 43
  Ethnicity Not Reported | 55 | 58 | 61 | 56 | 230
Body Mass Index in Kg/m^2 [Number; unit: participants]
  < 25 kg/m^2 | 3 | 6 | 10 | 7 | 26
  >=25 kg/m^2 | 65 | 66 | 64 | 61 | 256
  >=27 kg/m^2 | 60 | 57 | 54 | 48 | 219
  >=30 kg/m^2 | 41 | 48 | 45 | 37 | 171
Hemoglobin A1c (HbA1c) % [Mean (Standard Deviation); unit: Percent of Hemoglobin] | 7.80 (1.117) | 7.80 (0.984) | 8.11 (1.072) | 7.94 (1.029) | 7.92 (1.054)
Waist Circumference [Mean (Standard Deviation); unit: cm] — Waist was measured in centimeters (cm).
  cm | 105.24 (12.653) | 104.14 (11.642) | 101.48 (12.710) | 103.29 (13.745) | 103.50 (12.703)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1c (HbA1c) at Week 24 Last Observation Carried Forward (LOCF) - All Randomized Participants
Description: Adjusted mean change in HbA1c from baseline at Week 24, or the last post-baseline measurement prior to Week 24 if no Week 24 assessment was available was determined(LOCF). HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication (metformin) was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c values were obtained at enrollment, lead-in, and at Day 1, Weeks 4, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: Baseline (Day 1), Week 24
Population: N= Number of randomized participants, who took at least 1 dose of double-blind study medication, with non missing baseline and Week 24 (LOCF) values.
Measure: Mean (Standard Error); unit: Percent Hemoglobin
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Number analyzed (Participants) | 68 | 72 | 72 | 66
Percent Hemoglobin | 0.02 (0.1200) [-0.22 to 0.25] | -0.68 (0.1166) [-0.91 to -0.45] | -0.72 (0.1169) [-0.95 to -0.49] | -0.82 (0.1217) [-1.06 to -0.58]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 1mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Tested at alpha=0.019 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.02 to -0.37], Standard Error of Mean 0.1672
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 2.5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Tested at alpha=0.019 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.07 to -0.41], Standard Error of Mean 0.1679
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Tested at alpha=0.019 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.17 to -0.50], Standard Error of Mean 0.1710

2. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight at Week 24 (LOCF) - Randomized Participants
Description: Adjusted mean change in total body weight from baseline at Week 24, or the last post-baseline measurement prior to Week 24 if no Week 24 assessment was available LOCF was determined. Data after rescue medication (metformin) was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight was measured in kilograms (kg) at qualification, lead-in, Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, and 24 during double-blind period.
Time Frame: Baseline (Day 1), Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Number analyzed (Participants) | 68 | 72 | 74 | 67
kg | -0.96 (0.3942) | -2.69 (0.3820) | -2.64 (0.3776) | -2.69 (0.3961)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 1mg; By applying sequential testing procedure, the testing was performed since the primary endpoint was significant; Test type: Superiority or Other; p = 0.0018, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-2.81 to -0.65], Standard Error of Mean 0.5481
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 2.5 mg; Test type: Superiority or Other; p = 0.0024, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -1.68, 95% CI 2-sided [-2.76 to -0.60], Standard Error of Mean 0.5474
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p = 0.0022, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-2.83 to -0.63], Standard Error of Mean 0.5598

3. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose at Week 24 (LOCF) - Randomized Participants
Description: Adjusted mean change in fasting plasma glucose (FPG) from baseline at Week 24 (LOCF) was determined. Data after rescue medication (metformin) was excluded from this analysis. FPG was measured as milligrams per deciliter (mg/dL) by a central laboratory at qualification, lead-in, Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, and 24 during double-blind period. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: Baseline (Day 1), Week 24
Population: Number analyzed = Number of randomized participants, who took at least 1 dose of double-blind study medication, with non missing baseline and Week 24 (LOCF) values.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Number analyzed (Participants) | 68 | 72 | 74 | 67
mg/dL | 4.1 (4.200) | -11.0 (4.082) | -21.6 (4.025) | -28.5 (4.230)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 1mg; Test type: Superiority or Other; p = 0.0103, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -15.1, 95% CI 2-sided [-26.7 to -3.6], Standard Error of Mean 5.859
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 2.5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -25.7, 95% CI 2-sided [-37.2 to -14.3], Standard Error of Mean 5.816
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -32.6, 95% CI 2-sided [-44.3 to -20.8], Standard Error of Mean 5.962

4. Secondary Outcome: Adjusted Mean Change From Baseline in Effect on 2-hour Post Liquid Meal Glucose at Week 24 (LOCF) - Randomized Participants
Description: Liquid meal tolerance tests (MTTs) were scheduled to occur at Day 1 visit (MTT was to be completed 2 hours prior to first dose of treatment) and at Week 24 / End of treatment visit, or Rescue visit for participants meeting criteria for rescue due to lack of glycemic control. At Week 24, study treatment was given 1 hour before MTT was administered. Participant fasted for at least 10 hours (h) prior to both visits and abstained from tobacco, alcohol, and caffeine for 24 h prior to the MTT. The liquid meal supplement was administered over 10 minutes, starting immediately after Time 0 blood sample was drawn. Blood samples for post-liquid meal Glucose were obtained at 30, 60, 120, and 180 minutes after ingesting the liquid supplement. Glucose was measured in milligrams per deciliter (mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of double-blind study medication.
Time Frame: Baseline (Day 1), Week 24
Population: Number of randomized participants, who took at least 1 dose of double-blind study medication, with non missing baseline and Week 24 (LOCF) values.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Number analyzed (Participants) | 58 | 67 | 58 | 58
mg/dL | 8.81 (6.4925) | -33.3 (6.0390) | -39.3 (6.5025) | -51.8 (6.4973)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 1mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -42.1, 95% CI 2-sided [-59.56 to -24.61], Standard Error of Mean 8.8681
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 2.5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -48.1, 95% CI 2-sided [-66.27 to -30.03], Standard Error of Mean 9.1963
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 5 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -60.6, 95% CI 2-sided [-78.67 to -42.50], Standard Error of Mean 9.1796

5. Secondary Outcome: Adjusted Percentage of Participants Achieving a Therapeutic Glycemic Response at Week 24 (LOCF) - Randomized Participants
Description: Therapeutic glycemic response was defined as HbA1c less than 7.0%. n=Number of participants with HBA1c less than (<) 7 % at Week 24, last observation carried forward (LOCF) while N=number of randomized participants with non-missing baseline and Week 24 (LOCF) values. Percent=n/N and was adjusted for Baseline HbA1c. Data after rescue medication (metformin) was excluded from this analysis. HbA1c was measured as a percent of hemoglobin.
Time Frame: Baseline (Day 1), Week 24
Population: N=number of randomized participants with non-missing baseline and Week 24 (LOCF) values.
Measure: Number; unit: Adjusted Percentage of participants
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Number analyzed (Participants) | 68 | 72 | 72 | 66
Adjusted Percentage of participants | 34.6 | 53.6 | 43.4 | 49.1
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 1mg; The probability of response was modeled using a logistic regression model with baseline HbA1c as the covariate. Treatment group estimates of response rate were then obtained by integrating each group's modeled probability of response over the observed distribution of baseline covariate (combined across groups); Test type: Superiority or Other; p = 0.0157, Regression, Logistic — Test was performed at alpha=0.05; Logistic regression based on the methodology of Zhang, Tsiatis and Davidian and Tsiatis, Davidian, Zhang and Lu, with adjustment for baseline HbA1c; percent difference = 18.9, 95% CI 2-sided [3.6 to 34.3], Standard Error of Mean 7.380
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 2.5 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2512, Regression, Logistic — Test was performed at alpha=0.05; [statistical method as in outcome 5, analysis 1]; Percent Difference = 8.8, 95% CI 2-sided [-6.2 to 23.8], Standard Error of Mean 7.650
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 5 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0726, Regression, Logistic — Test was performed at alpha=0.05; [statistical method as in outcome 5, analysis 1]; Percent Difference = 14.5, 95% CI 2-sided [-1.3 to 30.3], Standard Error of Mean 8.069

6. Secondary Outcome: Adjusted Mean Change From Baseline in Waist Circumference at Week 24 (LOCF) - Randomization Participants
Description: Adjusted mean waist circumference values from baseline to Week 24 (or the last post-baseline measurement prior to Week 24 if no Week 24 assessment was available, last observation carried forward, (LOCF) was determined. Data after rescue medication (metformin) was excluded from this analysis. Waist circumference was measured centimeters (cm) and obtained at lead-in, Day 1, and Week 24 of the double-blind period. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: Baseline (Day 1), Week 24
Population: as for outcome 4
Measure: Mean (Standard Error); unit: cm
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Number analyzed (Participants) | 66 | 70 | 65 | 61
cm | -1.70 (0.5718) | -2.50 (0.5540) | -2.31 (0.5775) | -3.17 (0.5933)
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin 1mg; Test type: Superiority or Other; p = 0.3163, ANCOVA — Test was performed at alpha=0.05; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-2.37 to 0.77], Standard Error of Mean 0.7954
Statistical Analysis 2: Comparison: Placebo vs Dapagliflozin 2.5 mg; Following a sequential testing procedure, this comparison was not statistically tested, ie, the previous comparison did not meet the criterion for statistical significance; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-2.22 to 0.99], Standard Error of Mean 0.8154
Statistical Analysis 3: Comparison: Placebo vs Dapagliflozin 5 mg; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-3.09 to 0.16], Standard Error of Mean 0.8238

7. Secondary Outcome: Number of Participants With Deaths, Serious AEs (SAEs), Adverse Events (AEs), Discontinuation Due to AEs, During the 12 Week Double Blind Period, Including Data After Rescue - All Treated Participants
Description: Medical Dictionary for Regulatory Activities (MedDRA), version 12.1 AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug as per the investigator. Baseline to last dose plus 4 days for AEs, plus 30 days for SAEs. Data after rescue included.
Time Frame: Day 1 of Double Blind Period to end of Week 24 Plus 30 days
Population: Participants who received at least 1 dose of double-blind study medication during the double-blind treatment period. Data after rescue were also included.
Measure: Number; unit: participants
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Number analyzed (Participants) | 68 | 72 | 74 | 68
participants
  Death | 0 | 0 | 0 | 0
  Serious Adverse Event (SAE) | 0 | 2 | 2 | 0
  Related SAE | 0 | 2 | 0 | 0
  Adverse Event (AE) | 41 | 42 | 43 | 39
  Related Adverse Event | 8 | 5 | 9 | 5
  Discontinued due to AE | 0 | 1 | 1 | 0

8. Secondary Outcome: Number of Participants With Adverse Events of Special Interest During the 12 Week Double Blind Period - All Treated Participants
Description: Participants with AEs of hypoglycemia, cardiac/vascular disorders, renal impairment or failure, volume depletion (hypotension/dehydration/hypovolemia), fractures, urinary stones, and other reports suggestive of genital infection or urinary tract infection (UTI) were summarized using MedDRA version 12.1. Data after rescue included for all AEs of special interest except hypoglycemia; hypoglycemia AEs were prior to rescue. Major hypoglycemic episode: symptomatic requiring 3rd party assistance due to severe impairment in consciousness or behavior with a glucose value < 54 mg/dL and prompt recovery after glucose/glucagon; Minor: either symptomatic with glucose measurement < 63 mg/dL, regardless of need for 3rd party assistance, or asymptomatic with glucose < 63 mg/dL that does not qualify as major; Other: suggestive but not meeting criteria for major or minor.
Time Frame: Baseline to last dose plus 4 days in 12 Week Double Blind Period
Population: Randomized participants who received at least one dose of study medication in the double-blind period. Data after rescue included for all AEs of special interest except hypoglycemia; hypoglycemia AEs summarized below were prior to rescue.
Measure: Number; unit: participants
Groups:
- 1mg Dapagliflozin: 1 mg dapagliflozin tablets were taken orally once daily (with morning meal) for 24 weeks during the Double Blind Treatment Period.
- 2.5 mg Dapagliflozin: 2.5 mg dapagliflozin tablets were taken orally once daily (with morning meal) for 24 weeks during the Double Blind Treatment Period.
- 5 mg Dapagliflozin: 5 mg dapagliflozin tablets were taken orally once daily (with morning meal) for 24 weeks during the Double Blind Treatment Period.
Arm/Group | Placebo | 1mg Dapagliflozin | 2.5 mg Dapagliflozin | 5 mg Dapagliflozin
Number analyzed (Participants) | 68 | 72 | 74 | 68
participants
  Cardiac Disorders AEs | 0 | 0 | 4 | 0
  Vascular Disorders AEs | 4 | 1 | 2 | 1
  Hypoglycemia AEs (excluding data after rescue) | 0 | 0 | 1 | 1
  Major hypoglycemic episode | 0 | 0 | 0 | 0
  Minor hypoglycemic episode | 0 | 0 | 0 | 0
  Other hypoglycemic episode | 0 | 0 | 1 | 1
  AE Suggestive of Genital Infection | 2 | 1 | 5 | 2
  AE Suggestive of UTI | 1 | 3 | 1 | 2
  AE of Renal Impairment (creatinine increased) | 2 | 0 | 0 | 0
  AE of Hypotension | 0 | 0 | 0 | 1
  AE of Fracture | 3 | 0 | 0 | 0
  AE of Urinary Stones | 1 | 0 | 1 | 0

9. Secondary Outcome: Mean Change From Baseline in Seated Systolic and Diastolic Blood Pressure at Week 24, Including Data After Rescue - Treated Participants
Description: Blood pressure values were obtained on Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, and 24 in the double blind period, after the participant was seated for quietly for 5 minutes; the same arm (right or left) was used consistently through out the study. Measurements were taken at least 10 hours after the last ingestion of caffeine, alcohol, or nicotine. Blood pressure was measured in millimeters of mercury (mmHg). Data after rescue were also included. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: Baseline (Day 1), Week 24
Population: Participants who took at least 1 dose of double-blind study medication were analyzed. n= number of treated participants with non-missing baseline and Week 24 values.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg
Number analyzed (Participants) | 65 | 68 | 65 | 62
mmHg
  Systolic Blood Pressure (n=65, 68, 65, 62) | 0.8 (1.462) | -3.7 (1.449) | -3.1 (1.603) | -4.6 (1.531)
  Diastolic Blood Pressure (n=65, 68, 65, 62) | 0.2 (0.981) | -1.1 (1.040) | -2.0 (0.980) | -1.9 (1.036)

10. Secondary Outcome: Mean Change From Baseline in Seated Heart Rate at Week 24 - Treated Participants
Description: Heart rate values were obtained after the participant was seated for quietly for 5 minutes; the same arm (right or left) was used consistently through out the study. Measurements were taken at least 10 hours after the last ingestion of caffeine, alcohol, or nicotine. Heart rate was measured in beats per minute (bpm). Data after rescue were also included. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication.
Time Frame: Baseline (Day 1), Week 24
Population: N=number of participants who took at least 1 dose of double-blind study medication, with non missing baseline and Week 24 values.
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Placebo | 1mg Dapagliflozin | 2.5 mg Dapagliflozin | 5 mg Dapagliflozin
Number analyzed (Participants) | 65 | 68 | 65 | 62
bpm | -1.3 (1.178) | -2.0 (0.882) | -1.6 (0.845) | -1.4 (1.080)

11. Secondary Outcome: Number of Participants With Normal or Abnormal Electrocardiogram Summary Tracing at Week 24 (LOCF) - Treated Participants
Description: 12-Lead electrocardiograms (ECGs) were performed at Day -14 and Week 24/End of treatment visit (last observation carried forward) on participants who were supine. ECGs were assessed by the investigator. Baseline (BL) was Day -14 for this parameter.
Time Frame: Week 24
Population: N= Number of randomized participants, who took at least 1 dose of double-blind study medication, with non missing baseline (BL) and Week 24 (LOCF) values.
Measure: Number; unit: participants
Arm/Group | Placebo | 1mg Dapagliflozin | 2.5 mg Dapagliflozin | 5 mg Dapagliflozin
Number analyzed (Participants) | 68 | 72 | 74 | 68
participants
  Normal at BL, Normal at Week 24 (N=68, 72, 74, 68) | 34 | 38 | 43 | 38
  Abnormal BL, Normal at Week 24(N=68, 72, 74, 68) | 10 | 5 | 4 | 7
  Normal BL, Abnormal at Week 24(N=68, 72, 74, 68) | 4 | 3 | 4 | 1
  Abnormal BL, Abnormal at Week 24(N=68, 72, 74, 68) | 16 | 23 | 14 | 16
  Reported at BL, Not Reported at Week 24 | 4 | 3 | 9 | 6

12. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities in 24 Week Double Blind Treatment Period - Treated Participants
Description: Safety laboratory measurements were obtained at Day 1, Weeks 1, 2, 4, 8, 12, 20, and 24 in the double blind Period. Baseline was defined as the last assessment prior to the start of the first dose of the double-blind study medication. Data included from baseline up to and including the last day of treatment plus 4 days. Data after rescue was also included. Abbreviations; Pretreatment (PreRX); grams per deciliter (g/dL); upper limit of normal (ULN); milliequivalent per liter (mEq/L); greater than (>) less than (<); Units per liter (U/L), alanine aminotransferase (ALT); aspartate aminotransferase (AST); alkaline phosphatase (ALP); blood urea nitrogen (BUN). Marked abnormality Low (High) defined: hemoglobin <6 (>18 females or >20 males) g/dL; hematocrit <20% ( >55% females or >60% males); BUN (>60 mg/dL) or Urea >21.4 mmol/L; creatinine (>=1.5*preRX, >=2.5 mg/dL); AST and ALT >3*ULN; bilirubin >1.5*ULN; ALP >1.5*ULN.
Time Frame: Baseline to Week 24/end of treatment plus 4 days
Population: N=Number of participants who received at least 1 dose of study medication and had non-missing laboratory results.
Measure: Number; unit: participants
Arm/Group | Placebo | 1mg Dapagliflozin | 2.5 mg Dapagliflozin | 5 mg Dapagliflozin
Number analyzed (Participants) | 68 | 72 | 74 | 67
participants
  Hematocrit High >55% (N=68, 72, 74, 67) | 0 | 0 | 1 | 0
  Hemoglobin High >18 g/dL(N=68, 72, 74, 67) | 1 | 1 | 1 | 1
  Creatinine High >=1.5*PreRX(N=68, 72, 74, 67) | 2 | 1 | 1 | 4
  AST 3*ULN (N=68, 72, 74, 67) | 1 | 1 | 0 | 0
  ALT 3*ULN (N=68, 72, 74, 67) | 1 | 1 | 0 | 0
  ALT 5*ULN (N=68, 72, 74, 67) | 1 | 1 | 0 | 0
  AST or ALT >3*ULN (N=68, 72, 74, 67) | 1 | 1 | 0 | 0
  AST or ALT >5*ULN (N=68, 72, 74, 67) | 1 | 1 | 0 | 0
  Total bilirubin >1.5*ULN (N=68, 72, 74, 67) | 2 | 0 | 1 | 0
  Total bilirubin >2*ULN (N=68, 72, 74, 67) | 1 | 0 | 0 | 0
  ALP >1.5*ULN (N=68, 72, 74, 67) | 1 | 3 | 1 | 1
  ALP >3*ULN (N=68, 72, 74, 67) | 1 | 0 | 0 | 0
  Glucose >350 mg/dL (N=68, 72, 74, 67) | 1 | 1 | 0 | 0
  Creatinine Kinase > 5X ULN (N=68, 72, 74, 67) | 0 | 3 | 0 | 0
  Calcium <7.5 mg/dL (N=68, 72, 74, 67) | 1 | 2 | 0 | 0
  Calcium (mg/dL) >=1 vs ULN and >=0.5 vs baseline | 1 | 0 | 0 | 0
  Potassium >= 6 meq/L (N=68, 72, 74, 67) | 0 | 0 | 2 | 1
  Magnesium <1 meq/L (N=68, 72, 74, 67) | 1 | 1 | 0 | 0
  Sodium <130 meq/L (N=68, 72, 74, 67) | 1 | 1 | 0 | 0
  Sodium >150 meq/L (N=68, 72, 74, 67) | 0 | 0 | 1 | 0
  Sodium < 120 meq/L | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 Weeks plus 30 days; Day 1 of double blind treatment to last patient, last visit.
Arm/Group | Dapagliflozin 1mg | Dapagliflozin 2.5 mg | Dapagliflozin 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/72 | 2/74 | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 14/72 | 14/74 | 7/68 | 18/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 1mg (N=72) | Dapagliflozin 2.5 mg (N=74) | Dapagliflozin 5 mg (N=68) | Placebo (N=68)
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 1mg (N=72) | Dapagliflozin 2.5 mg (N=74) | Dapagliflozin 5 mg (N=68) | Placebo (N=68)
Headache (Nervous system disorders) | 5 | 4 | 2 | 5
Pharyngitis (Infections and infestations) | 1 | 4 | 2 | 3
Nasopharyngitis (Infections and infestations) | 5 | 1 | 2 | 3
Dizziness (Nervous system disorders) | 3 | 5 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.